CLINICAL TRIAL: NCT06188533
Title: Urinary Activin A as Apredictive Marker for Assessement of Acute Kidney Injury Severity in Patient Admitted at Assuit University Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kamal mahmoud mohamed amin, Principal investigator, Assiut University
Other Study IDs: Urinary activin A in AKI
Record Dates: First submitted 2023-12-19; First posted 2024-01-03 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Urinary Activin A in AKI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Urinary activin A in AKI — Urinary activin A in AKI patient

SUMMARY:
Urinary Activin A as amarker for assessement of acute kidney injury severity in patient admitted at Assuit University Hospital

DETAILED DESCRIPTION:
Acute kidney injury has been ahealth problem all over the world , It's prevelance in developing and developed countries is increasing due to pre renal , renal , post renal causes .

Estimates of AKI prevalence range from <1% to 66%. These variations can be explained by not only population differences but also inconsistent use of standardized AKI classification criteria. The aetiology and incidence of AKI also differ between high-income and low-to-middle-income countries.(1)

* It can be presented in different stages according to AKIN classification (stage l (Increase in serum creatinine ≥0.3md/dl (≥26.4μmol/l) or increase to >150% to 200% (1.5 fold to 2 fold) from baseline , and urine output (<0.5 ml/kg/h for >6 h ))

  * stage ll (Increase to >200% to 300% (>2 fold to 3 fold) from baseline) , and urine output (<0.5 ml/kg/h for >12 h ))
  * stage lll(Increase in serum creatinine to >300% (>3 fold) from baseline, or serum creatinine >4.0mg/dl (>354μmol/l) with acute increase of atleast 0.5mg/dl ) Urine output(<0.3ml/kg/hr for 24 hours, or anuria for 12 hours). (2)
* In ischemic kidney, there is acytokine belong to the transforming growth factor (TGF)-B ( Activin A) that regulates the growth and differantiation of cell in variuos organs was significantly increasd in ischemic kidney . (3)
* level of Activin A in urine correlate to the severity of the acute kidney injury (AKI), as the level of urinary Activin A in first stages of acute kidney injury is less than the second and third stages . (4)
* so follow up of urinary Activin A in patients with acute kidney injury can be avery useful biomarker for assessement of severity of acute kidney injury. (4)

ELIGIBILITY:
Inclusion Criteria:

* The study will include patient with acute kidney injury with no history of chronic kidney diseases

Exclusion Criteria:

* patient with history of chronic kidney diseases , diseases associated with icreased activin A level such as ( heart failure , cancers , COPD , systemic sclerosis ,pregnant , viral infection , and Mycosis Fungoides and Sézary Syndrom

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * level of Activin A in urine correlate to the severity of the acute kidney injury (AKI), as the level of urinary Activin A in first stages of acute kidney injury is less than the second and third stages . (4)
  * so follow up of urinary Activin A in patients with acute kidney injury can be avery useful biomarker for assessement of severity of acute kidney injury
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Urinary activin A in AKI | Baseline
  To correlate between Activin A level in urine and severity of AKI